CLINICAL TRIAL: NCT02964637
Title: Multimodal Assessment for Predicting Specific Pathological Substrate in Frontotemporal Lobar Degeneration
Brief Title: Diagnosing Frontotemporal Lobar Degeneration
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, Principal Investigator, University Health Network, Toronto
Other Study IDs: 14-8398-A
Record Dates: First submitted 2016-09-23; First posted 2016-11-16 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2019-04

CONDITIONS: Corticobasal Syndrome; Progressive Supranuclear Palsy; Behavioral Variant Frontotemporal Dementia; Semantic Dementia; Progressive Nonfluent Aphasia; Amyotrophic Lateral Sclerosis And/or Frontotemporal Dementia
MeSH Terms: conditions — Corticobasal Degeneration; Supranuclear Palsy, Progressive; Frontotemporal Dementia; Primary Progressive Nonfluent Aphasia; Frontotemporal Dementia With Motor Neuron Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood for biomarkers will be collected from participants for genetic testing. In addition, cerebrospinal fluid (CSF) will be collected to measure levels of different proteins, such as tau.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Progressive supranuclear palsy: Observational Study
  Interventions: Other: Observational Study
- Corticobasal syndrome: Observational Study
  Interventions: Other: Observational Study
- Behavoral variant FTD: Observational Study
  Interventions: Other: Observational Study
- Semantic variant PPA: Observational Study
  Interventions: Other: Observational Study
- Non-fluent variant PPA: Observational Study
  Interventions: Other: Observational Study
- FTD-motor neuron disease: Observational Study
  Interventions: Other: Observational Study
- Healthy controls: Observational Study
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study

SUMMARY:
To establish diagnostic tools to make an accurate clinical and pathological diagnosis of patients with clinical FTLD syndromes

DETAILED DESCRIPTION:
The goal of this study is to determine the best diagnostic test for diagnosing frontotemporal lobar degeneration. To accomplish this, the current study will evaluate different tests: brain imaging, skin biopsy, body fluid samples (blood and cerebrospinal fluid), thinking abilities, everyday functioning, and brain autopsy. The study team hopes that this information can be used to guide diagnosis and further understanding of mechanism of disease in Frontotemporal Lobar Degeneration and possibly treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a reliable study partner who can provide an independent evaluation of functioning.
* Able to read, understand and speak English for neuropsychological testing.
* All subjects must meet one of these diagnostic criteria (A) probable behavioral variant FTD, (B) MRI-supported non-fluent variant PPA; (C) MRI-supported semantic variant PPA and [18F]T807 negative (D) probable CBS: using current criteria for CBS(27); (E) PSP: inclusion criteria for PSP are based upon the National Institute of Neurological Disorders and Stroke Society of Progressive Supranuclear Palsy (NINDS-SPSP) (F) FTD-MND
* Control subjects must have a normal neurological exam, a CDR sum of boxes = 0, and MMSE score equal to or greater than 28

Exclusion Criteria:

* Patients with clinical, imaging or CSF A beta/ tau profile consistent with AD
* History of traumatic brain injury, brain tumors, stroke or other neurological or psychiatric disorders that can explain symptoms will be excluded.
* Premenopausal women will be asked to consent to a pregnancy test prior to each scan as pregnant women will be excluded from study because of potential harm to fetus from PET study.
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of progressive supranuclear palsy (PSP), corticobasal syndrome (CBS), semantic variant primary progressive aphasia (sv-PPA), non-fluent variant PPA (nfv-PPA), behavioral variant frontotemporal dementia (bvFTD) or FTD-motor neuron disease (FTD-MND).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Structural and Functional Diffferences between the FTLD groups via MRI of the brain | One time visit through study completion of 5 years
  Differences in brain volumes and resting state functional connectivity
Differences between the FTLD groups via PET imaging of the brain | One time visit through study completion of 5 years
  Differences in ligand uptake

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Tartaglia, M.D., Principal Investigator — Toronto Western Hospital, UHN; Tanz CRND
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No